CLINICAL TRIAL: NCT04966169
Title: Effectiveness of GentleWave on the Healing of Apical Periodontitis: A Prospective Cohort Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Departure from the University of Iowa
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202102255
Record Dates: First submitted 2021-07-07; First posted 2021-07-19 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sonendo GentleWave (Experimental): Every participant will receive the same experimental treatment, which is root canal therapy using the Sonendo GentleWave System.
  Interventions: Device: GentleWave System

INTERVENTIONS:
Device: GentleWave System — The GentleWave hydrodynamic cavitation system is a 510k FDA-approved multisonic energy system that is used in complex root canal procedures.

SUMMARY:
The purpose of this 12-month prospective cohort study is to evaluate post-operatory pain, patient satisfaction, and treatment outcomes (i.e., healing) when the newly-developed, 510k FDA-approved multisonic energy GentleWAve System (Sonendo, Inc., Laguna Hills, CA) is used in complex root canal procedures.

DETAILED DESCRIPTION:
Apical Periodontitis (AP) is a disease where multiple types of bacteria, including those that can live without oxygen, create a bacterial film on the tissues around teeth. These bacteria colonize the dying pulp tissue, invade channels within teeth and other openings, and create an inflammatory response of the tissues surrounding the teeth. Therefore, the primary goal of endodontic treatment is to reduce bacteria numbers by removing remaining tissues, bacterial films, and infected dentine (i.e., layer of tooth below the enamel). Healing of apical periodontitis (AP) is expected, in the majority of cases, if proper bacterial disinfection is accomplished.

Elimination of these bacteria can be achieved by a combined action of several treatments. Lately, irrigation and mechanical instrumentation techniques have been developed with this intention. Some new technologies are based on the concept of using minimally-invasive instruments with hydrodynamic cavitation generating a broad spectrum of sound waves within the degassed fluid inside of the tooth. However, there is not enough evidence in the literature to support its efficacy.

The hypothesis of this study is that the GentleWave (GW) hydrodynamic cavitation system (Sonendo, Inc., Laguna Hills, CA) will achieve a high success rate in treating and healing apical periodontitis (AP), a disease where a bacterial film is formed on the tissues around the teeth.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years
* Speak and Read English
* Able to attend follow-up visits at 6 months AND 1 year (post-baseline treatment)
* A tooth with no response to cold and electric pulp testing.
* Tooth is a 1st or 2nd mandibular molar
* Tooth has no response to cold/electric pulp testing
* Tooth has a diagnosis of pulp necrosis with asymptomatic apical periodontitis
* 1st and 2nd mandibular molars.
* Current (i.e., taken within the last week) radiograph available (or done at screening, as needed)
* A limited-volume, cone-beam computed tomography (CBCT) taken at the first visit confirms apical periodontitis (radiolucency).

Exclusion Criteria:

* Patient has advanced untreated periodontal disease/recent periodontal surgery
* Patient has non-odontogenic facial pan (e.g., face pain of unknown cause)
* Patient has a history of poor attendance at dental visits
* Patient is pregnant
* Patient reports taking corticosteroids
* Patient is supervised by the Principal Investigator or a member of the research team
* Patient is subordinate to the Principal Investigator or a member of the research team
* Patient is a student/trainee under the direction of the Principal Investigator or a member of the research team
* Tooth had previous intervention (e.g., pulp debridement: removal of the pulp/nerve of the tooth)
* Tooth has incomplete root formation (e.g., immature with apical periodontitis)
* Tooth has defective restorations or carious lesions (i.e., cavities) that could lead to microleakage
* Tooth has internal or external resorption
* Tooth has a mobility score of 3
* Tooth has a fracture/visibly cracked
* Tooth has vital (i.e., functioning) pulp
* Advanced untreated periodontal disease or recent periodontal surgery.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Cone Beam Computed Tomography Periapical Index (CBCTPAI) across 1 year | Baseline; 6-months; 12 months
  This will be assessed by the evaluator measuring the estimated tooth on the CBCT and assigning an index score on the CBCT. A score of 0 denotes an intact periapical bone structure. A score of 1 denotes a diameter of periapical radiolucency >0.5-1mm. A score of 2 denotes a diameter of periapical radiolucency >1-2mm. A score of 3 denotes a diameter of periapical radiolucency >2-4mm. A score of 4 denotes a diameter of periapical radiolucency >4-8mm. A score of 5 denotes a diameter of periapical radiolucency >8mm. A score of 6 denotes (n) + E = expansion of periapical cortical bone. A score of 7 denotes (n) + D = destruction of periapical cortical bone.
Change from baseline of peripical index (PAI) across 1 year. | Baseline; 6-months post-baseline; 12 months post-baseline
  This will be assessed by asking the evaluator to evaluate the PAI score at each X-ray. A value of 1 denotes normal periapical structures. A value of 2 denotes small changes in the bone structure. A value of 3 denotes changes in bone structure with some mineral loss. A value of 4 denotes apical periodontitis with well-defined radiolucent areas. A value of 5 denotes severe apical periodontitis with exacerbating features.
Change from baseline of modified wound healing scale (Mod-CWHS) across 1 year | 6 months post-baseline; 12 months post-baseline
  This will be assessed by the evaluator evaluating the research subject's healing status on a scale of 1-3. A value of 1 is "Uneventful wound healing with no gingival edema, erythema, suppuration, discomfort or barrier exposure. A value of 2 is "Uneventful wound healing with slight gingival edema, erythema, or discomfort but no suppuration. 3 is a value of poor wound healing with significant gingival edema, erythema, discomfort, loss of barrier or any suppuration.
Change from baseline of pain severity in 0-10 pain severity scale across 1 year | Baseline; 2 days post-baseline; 1 weeks post-baseline; 2 weeks post-baseline; 6 months post-baseline; 12-months post-baseline
  This will be assessed by asking the research subject their current level of pain on a 0-10 scale, and the patient will circle one line.
Change from Day 2 of research subject's thoughts on treatment result across 1 year. | 2 days post-baseline; 1-week post-baseline; 2-weeks post-baseline; 6-months post-baseline; 12 months post-baseline
  This will be assessed by asking the research subject to assess their own treatment result on a scale of 0 to 10 and circling one line.

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio Teixeira, DDS,MS,PhD, Principal Investigator — University of Iowa College of Dentistry
Locations (1):
- University of Iowa College of Dentistry and Dental Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grigsby D Jr, Ordinola-Zapata R, McClanahan SB, Fok A. Postoperative Pain after Treatment Using the GentleWave System: A Randomized Controlled Trial. J Endod. 2020 Aug;46(8):1017-1022. doi: 10.1016/j.joen.2020.04.004. Epub 2020 Jun 14. PMID 32553417
- [Background] Sigurdsson A, Le KT, Woo SM, Rassoulian SA, McLachlan K, Abbassi F, Garland RW. Six-month healing success rates after endodontic treatment using the novel GentleWave System: The pure prospective multi-center clinical study. J Clin Exp Dent. 2016 Jul 1;8(3):e290-8. doi: 10.4317/jced.52779. eCollection 2016 Jul. PMID 27398180
- [Background] Sigurdsson A, Garland RW, Le KT, Woo SM. 12-month Healing Rates after Endodontic Therapy Using the Novel GentleWave System: A Prospective Multicenter Clinical Study. J Endod. 2016 Jul;42(7):1040-8. doi: 10.1016/j.joen.2016.04.017. PMID 27325455
- [Background] Wohlgemuth P, Cuocolo D, Vandrangi P, Sigurdsson A. Effectiveness of the GentleWave System in Removing Separated Instruments. J Endod. 2015 Nov;41(11):1895-8. doi: 10.1016/j.joen.2015.08.015. Epub 2015 Sep 26. PMID 26409807